CLINICAL TRIAL: NCT01228643
Title: Study Of Effectiveness Of The Use Of Pancreatic Enzyme: Norzyme® -(Made In The Laboratory Pancrealipase Bergamo) Inpatients With Pancreatic Insufficiency In Use Substituteenzymatic When Compared To Product Creon®
Brief Title: Effectiveness of Pancreatic Enzymes in Patients Pancreatic Insufficient: Comparison of Two Drugs
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Principal Investigator, Azidus Brasil, Principal Investigator Dr. Alexandre Frederico, Azidus Brasil
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PANBER0607
Record Dates: First submitted 2008-02-11; First posted 2010-10-26 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Chronic Renal Failure
Keywords: Pancreatic enzymes.; To evaluate the efficacy of drugs in chronic renal failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Norzyme® (Experimental)
  Interventions: Biological: Pancreatic enzimes
- Creon® (Active Comparator)
  Interventions: Device: Creon ®

INTERVENTIONS:
Biological: Pancreatic enzimes — - Norzyme ® (product testing) composition: 20.000USP lipase, 65.000USP of 65.000USP amylase and protease.
  Arms: Norzyme®
Device: Creon ® — - Creon ® (reference product) composition: 25.000UI lipase, amylase 74.700UI 62.500UI and protease
  Arms: Creon®

SUMMARY:
Prove the efficacy of pancreatic enzyme Norzyme ® imported by Pharmaceutical Chemistry Laboratory Bergamo Ltda. verified by activity lipase contained in the formulation in controlling steatorrhea in 16 patients of both sexes aged 14 to 65 years, patients with pancreatic insufficiency Exogenous any cause. It's effectiveness will be found in a study randomized, crossover, comparative biosimilar product produced by Creon ® Laboratory Solvay Farma Ltda.

DETAILED DESCRIPTION:
Phase III clinical trial systematic sampling, double-blind, randomized, crossed that evaluates the comparative efficacy of a formulation containing enzyme pancreas in 16 patients with pancreatic insufficiency exogenous of any cause. The study will be conducted with the inclusion of 16 adult patients, both sexes, regardless of color or social class, aged 14 to 65 years, clinically diagnosed as having pancreatic insufficiency exocrine any etiology (cystic fibrosis, cancer, pancreatectomy, Surgery by trauma). The Research Subjects will be recruited with the help of medical coinvestigador specialist Dr. Francisco Callejas Neto, who will offer their clinic patients to participate in the study. If there is interest from same, all are invited to attend the Clinic for total LAL clarification about the study of drug action, benefits, possible risks, compensation, study period, and finally understanding reading and signing together with the investigator of the Term of Consent.

The research subjects will have complete freedom to lead to the Informed Consent house, where they can review all items easy. After informed and the consent form and signed informed, patients will be examined by the researcher LAL Clinic which will perform a physical examination in the same general and specific. Will rated their personal background and reviewed the Inclusion and Excluded from the study.

Satisfying the criteria for inclusion in the study subjects are approved to participate in the study.

The 16 Subjects Research approved within the inclusion criteria and exclusion to participate in the study be included in the study as sequential by the number of their care. Later, the same will be inserted in randomization table, which was outlined in a randomized crossover for two drugs, the randomization scheme will be in the balanced cross 2 x 2. A design is said to be balanced if it satisfies the following conditions:

· Each medication is applied only once in each subject;

• in each period, the number of subjects receiving each medicine must be equal; This randomization was previously performed by the computer program and by a qualified professional Prof. Dr. Yuko Wada Cilicia (PhD in Biostatistics and PhD of Biostatistics, UNICAMP) of Statpharm Scientific Consulting Ltda.

All study medication will be labeled according to the randomization, previously performed by pharmacy LAL Clinica, which should make conference material for 3 checks. In each period of the study medication should be labeled with the following words: code of the subject during the study period and dose to be administered in the same. All these procedures should be made to minimize and avoid bias in the study.

ELIGIBILITY:
nclusion Criteria:

* Research subjects aged between 14 and 65 years of both sexes;
* Exogenous pancreatic insufficiency of any etiology;
* Subjects who do not regularly use or pancreatic enzymes by orally;
* Freely agree to sign the consent form and clarified before all the essential elements of the protocol be clarified before any procedure.

Exclusion Criteria:

* Participation in any study or have ingested some experimental drug trial in the 3 months preceding the study.
* Regular use of medication that interferes with the action of the drug test:
* in the 4 weeks preceding the study or make use of any medications that interfere with drug test a week before the start the study.
* Patients who take any kind of treatment for morbid obesity.
* Cases of stomach reduction surgery.
* Cases of surgical reduction of the intestine.
* Present history of current abuse of alcohol or have drunk alcohol in the 48 hours prior to the study.
* Have any condition which prevents him from participating in the study, for trial Principal Investigator.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Balance of fat in feces. | 06 weeks of treatment.

SECONDARY OUTCOMES:
Prove the efficacy of pancreatic enzyme Norzyme ® through the activity of lipase in the formulation contained in the control of steatorrhea | 06 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Frederico, Doctor, Principal Investigator — LAL Clinical Reseach e Development Ltda
Locations (1):
- LAL Clinica Pesquisa e Desenvolvimento LTDA, Valinhos, São Paulo, Brazil